CLINICAL TRIAL: NCT00009802
Title: A Phase I Trial Of Oral Calcitriol [1,25-(OH)2D3] And Paclitaxel In Advanced Solid Tumors
Brief Title: Calcitriol Plus Paclitaxel in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Laura A. Pollice, Clinical Research Manager, University of Pittsburgh
Purpose: Treatment
Other Study IDs: 98-019; CDR0000068411 (Registry Identifier: PDQ (Physician Data Query)); PCI-IRB-980542; NCI-G00-1901
Record Dates: First submitted 2001-02-02; First posted 2003-06-06 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Calcitriol; Paclitaxel

INTERVENTIONS:
Dietary Supplement: calcitriol
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Calcitriol may increase the effectiveness of paclitaxel by making tumor cells more sensitive to the drug.

PURPOSE: Phase I trial to study the effectiveness of combining calcitriol with paclitaxel in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxic effects and maximum tolerated dose of calcitriol when combined with paclitaxel in patients with advanced solid tumors.
* Determine the effect of administration of calcitriol on the pharmacokinetics of paclitaxel in these patients.
* Determine the effect of administration of paclitaxel on the pharmacokinetics of calcitriol in these patients.

OUTLINE: This is a dose-escalation study of calcitriol.

During course 1, patients receive oral calcitriol daily on days 1-3 of weeks 1-6 and paclitaxel IV over 1 hour on day 1 of week 1 and day 3 of weeks 2-6. During course 2 and subsequent courses, patients receive oral calcitriol daily on days 1-3 and paclitaxel IV over 1 hour on day 3 of weeks 1-6. Treatment continues every 8 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of calcitriol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the highest dose giving an estimated probability of dose-limiting toxicity of no more than 0.30.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven advanced cancer not curable by standard therapies
* Brain metastases allowed following definitive radiotherapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 4 times normal

Renal:

* Creatinine no greater than 2.0 mg/dL
* Calcium no greater than 10.5 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-barrier contraception for at least 1 week before, during, and for at least 2 weeks after study
* No active infection or serious concurrent condition
* No symptomatic peripheral neuropathy greater than grade 1

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior regional or systemic biologic therapy

Chemotherapy:

* At least 3 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosourea)

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 1998-06; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh K. Ramanathan, MD, Study Chair — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States